CLINICAL TRIAL: NCT04650971
Title: Phase I Randomized Double Blind Placebo-controlled Study of Universal Influenza Vector Vaccine "UniFluVec" of Two Dose Levels After Two Intranasal Administrations in Healthy Volunteers at the Age From 18 to 49 Years Old
Brief Title: Study to Assess Safety, Tolerability and Reactogenicity of Vaccine "UniFluVec" After Two Intranasal Administrations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmenterprises Biotech LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: UFV-I-01/2017
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Influenza A
Keywords: Healthy volunteers; Vector vaccine; UniFluVec

STUDY DESIGN:
Intervention Model Description: The dose cohorts were included into the study based on evaluation of the safety results performed by the Data Safety Monitoring Committee. 2 doses of vaccine/placebo were used in the study. The volunteers randomized to the study group received intranasally 0.5 ml of the vaccine/placebo (0.25 ml in each nostril) as nasal aerosol stray twice with an interval of 3 weeks.
Who Masked: Participant, Investigator
Masking Description: For blinding purposes the Placebo was made with the corresponding labelling of the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccine "UniFluVec" 6.7 log EID50/dose (Experimental): Cohort 1 - 30 subjects were randomized in a 2:1 ratio to be treated either with Vaccine "UniFluVec" 6.7 log EID50/dose (20 subjects) or with placebo (10 subject, see placebo arm).
  Interventions: Biological: UniFluVec
- Vaccine "UniFluVec" 7.7 log EID50/dose (Experimental): Cohort 2 - 30 subjects were randomized in a 2:1 ratio to be treated either with Vaccine "UniFluVec" 7.7 log EID50/dose (20 subjects) or with placebo (10 subject, see placebo arm).
  Interventions: Biological: UniFluVec
- Placebo (Placebo Comparator): Placebo comparator arm consists of 20 subjects (10 subject in each Сohort).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: UniFluVec — Vaccination was performed intranasally (0.25 ml in each nostril) twice with an interval of 3 weeks
  Arms: Vaccine "UniFluVec" 6.7 log EID50/dose; Vaccine "UniFluVec" 7.7 log EID50/dose
Biological: Placebo — Vaccination was performed intranasally (0.25 ml in each nostril) twice with an interval of 3 weeks
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled, Phase I clinical study of the safety, tolerability, reactogenicity and immunogenic activity of the universal influenza vector vaccine "UniFluVec" at two dose levels after two intranasal administrations in healthy adults. The volunteers randomized to the study group received intranasally 0.5 ml of the vaccine (0.25 ml in each nostril) as nasal aerosol stray twice with an interval of 3 weeks. The vaccine of the first dose level contained 6.7 log EID50/0.5 ml (50% egg infective dose) of attenuated recombinant influenza A/H1N1pdm09 virus; vaccine of the second dose level contained 7.7 log EID50/0.5 ml of attenuated recombinant influenza A/H1N1pdm09 virus.

The primary objective of the study was to evaluate the safety, tolerability and reactogenicity profile of vaccine "UniFluVec" based on the frequency and severity of adverse events. The secondary objective of the study was to assess the immunogenicity.

DETAILED DESCRIPTION:
One center located in Russia (Saint-Petersburg) was approved for participation in this study. The study consisted of 3 periods: screening, double vaccination with an interval of 3 weeks and follow-up.

All eligible subjects were randomized into the study in appropriate cohort groups sequentially. Randomization was performed within each cohort in ratio 2:1 to the vaccine and placebo groups, respectively:

* Cohort 1 (total 30 volunteers) - 20 volunteers received the vaccine twice, 6.7 log EID50/dose; 10 volunteers received Placebo twice.
* Cohort 2 (total 30 volunteers) - 20 volunteers received the vaccine twice, 7.7 log EID50/dose; 10 volunteers received Placebo twice.

The decision to administer the second dose of vaccine or increased vaccine dose (cohort 2) was approved by the Data Safety Monitoring Committee on the basis of preliminary safety results assessment.

The follow-up period lasted 3 months after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of signed informed consent.
2. Adult men and women at the age from 18 through 49 years old.
3. Diagnosis "healthy", verified by standard examination.
4. Body weight ≥ 50 kg.
5. The subjects, who are antibody-negative to influenza A/H1N1pdm virus (antibody titers ≤1:10 based on Hemagglutination inhibition assay (HIA)).
6. Ability and voluntary desire to keep records in the Self-Observation Diary, as well as to attend all the visits of the study for the medical control.
7. Consent of study subjects to use reliable contraception methods during the entire period of their participation in the study, as well as within 3 months after completion of participation in the study.

Exclusion Criteria:

1. Participation in another clinical study within three months prior to the beginning of this study; plans to participate in another study during the period of this study.
2. Immunization with any other vaccine, not provided by the study within 6 months prior to inclusion in this study, or refusal to postpone another immunization until the end of the four-week period after completion of this study.
3. Regular administration of irrigation therapy of the nasal cavity within the last six months prior to inclusion in this study or occasional application of this treatment method within two weeks prior to inclusion in this study.
4. Frequent nosebleeds within the year before the study in the past medical history (> 5).
5. Clinically significant anatomical pathology of the paranasal area or signs of surgical intervention in the area of the nose, sinus sinuses or traumatic injuries of the nose during the month before the beginning of screening.
6. Symptoms of acute respiratory disease, including fever, or other acute diseases as of the screening date or within two weeks before the beginning of screening.
7. Treatment with immunoglobulins or other blood products within three months prior to the beginning of screening or planning such treatment during participation in this study; blood/plasma donation (from 450 ml blood or plasma) in less than 2 months prior to screening.
8. The presence or suspicion of various immunosuppressive or immunodeficient conditions or continuous administration (the drug is prescribed for more than 14 days of continous administration) of immunosuppressive drugs, immunomodulators during 6 months before inclusion in this study (for corticosteroids - greater than or equal to 0.5 mg/kg of prednisolone or other equivalent corticosteroids per day; topical and inhaled steroids, except for administration in the nasal cavity, are allowed).
9. Participation in any previous studies to assess vaccines containing influenza viruses A/H1N1pdm09.
10. Severe allergic reactions, including asthma, Quincke's edema, anaphylactic shock in the past medical history.
11. Wheezing after a previous immunization with live influenza vaccine in the past medical history.
12. Hypersensitivity after any previous vaccination against influenza and/or adverse effects caused by immunization, like body temperature above 40°C, fainting, non-febrile convulsions, anaphylaxis, when there is a minimal risk of association with the previous administration of any vaccine (not only against influenza).
13. Suspected hypersensitivity to any components of the investigated vaccine, including chicken egg protein.
14. Seasonal (spring or autumn) hypersensitivity to the natural factor effects.
15. Acute or chronic clinically significant lesions in the lungs, the cardiovascular system, liver, endocrine, neurological and psychiatric diseases or renal dysfunction, as revealed based on the past medical history, physical examination or clinical laboratory findings, which may have an impact on the study results.
16. Leukemia or any other malignant blood diseases or solid malignant neoplasms of other organs in the past medical history.
17. Thrombocytopenic purpura blood-clotting disorders in the past medical history.
18. Seizures in the past medical history.
19. HIV, hepatitis B or C.
20. Tuberculosis.
21. Chronic alcohol addiction or chronic use of illegal drugs, drug abuse.
22. Pregnancy or breastfeeding.
23. Any condition that, according to the researcher, can increase the health risk for the volunteer participating in the study or influence the study results.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | Day -7 (7 days before first dose) - Day 111
  Adverse events (AEs) were summarized per treatment arm according to the current Medical Dictionary for Regulatory Activities (medDRA) version 21.1. For each preferred term, frequency counts and percentages were calculated.
  Related and unrelated AEs were assessed.
  Special attention was paid to vaccine-specific significant AEs:
  * Immediate AEs occurring within two hours after administration of the vaccine and detected both by the medical personnel and based on the information provided by the volunteer to the research staff.
  * Post-vaccination reactions (foreseen local and systemic clinical signs), usually caused by intranasal vaccination within two hours and the subsequent 7 days after administration of the vaccine.

SECONDARY OUTCOMES:
Assessment of the virus reisolation after the vaccination | Day 2 - Day 5, Day 23, Day 25
  This was evaluated according to the diagnostic rapid test for influenza A virus by immunochromatographic method in the nasal swab samples within control periods after vaccination
The content of serum antibodies | Day 1, Day 21, Day 42
  This was evaluated by Hemagglutinin-inhibition assay
The content of serum neutralizing antibodies | Day 1, Day 21, Day 42
  This was evaluated by microneutralization assay
The content of serum Immunoglobulins class G (IgG) | Day 1, Day 21, Day 42
  This was evaluated by enzyme-linked immunosorbent assay (ELISA)
The content of serum Immunoglobulins class E (IgE) | Day 1, Day 21, Day 42
  This was evaluated by ELISA
Determination of Myxovirus resistance (MxA) protein 1 | Day 1, Day 3 (1-st and 3-d days after first vaccination), Day 21, Day 23 (1th and 3th days after second vaccination)
  This was evaluated in the whole blood samples by ELISA
The content of secretory Immunoglobulins class A (IgA) and IgG | Day 1, Day 21, Day 42
  This was evaluated by ELISA and microneutralization assay in the samples of nasal secretions.

OTHER OUTCOMES:
The content of cytokines | Day 1, Day 2, Day 3
  This was evaluated by ELISA and detected in samples of nasal secretions

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution "Research Institute of Influenza" of the Ministry of Health of the Russian Federation, Saint Petersburg, Russia